CLINICAL TRIAL: NCT06469034
Title: Use of Head-mounted Display for Ultrasound-guided Central Venous Catheterization in Adults: a Randomized Controlled Study
Brief Title: Head-mounted Display for Central Venous Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Yun Wu, Doctor, Anesthesiology, Principal Investigator, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YX2024-066(F1)
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Central Venous Catheterization

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): The operators in the control group will perform the procedure by visualizing the conventional ultrasound images displayed directly on the ultrasound screen. Each operator will perform an internal jugular vein cannulation via the short-axis approach. To standardize the approach, the ultrasound machine will be placed just to the right of the patient and operators will be asked to stand at the head of the patient and perform the procedure on the patient's internal jugular vein. Each operator could determine the height of the surgical table, and the posture during the procedure that will be most familiar to him/her to increase the success rate. Every procedure will be recorded by focusing on the participant's hands and faces.
  Interventions: Device: conventional ultrasound
- HMD group (Experimental): In the HMD group, the ultrasound machine will be located behind the operator to remove the distraction, and the operator will not be allowed to see the ultrasound screen during the procedure. Images from the ultrasound will be transmitted to HMD via a novel connection developed specifically for this purpose. The operator will wear a pair of HMD and perform the procedure by visualizing the ultrasound images displayed on their HMD screen instead of the ultrasound screen. Each operator will perform an internal jugular vein cannulation via the short-axis approach. Every procedure will be recorded by focusing on the participant's hands and faces.
  Interventions: Device: Head-mounted display ultrasound

INTERVENTIONS:
Device: conventional ultrasound — The operators in the control group will perform the procedure by visualizing the conventional ultrasound images displayed directly on the ultrasound screen. Each operator will perform an internal jugular vein cannulation via the short-axis approach. To standardize the approach, the ultrasound machine will be placed just to the right of the patient and operators will be asked to stand at the head of the patient and perform the procedure on the patient's internal jugular vein. Each operator could determine the height of the surgical table, and the posture during the procedure that will be most familiar to him/her to increase the success rate. Every procedure will be recorded by focusing on the participant's hands and faces.
  Arms: Control group
Device: Head-mounted display ultrasound — In the HMD group, the ultrasound machine will be located behind the operator to remove the distraction, and the operator will not be allowed to see the ultrasound screen during the procedure. Images from the MR ultrasound machine will be transmitted to HMD via a novel connection developed specifically for this purpose. The operator will wear a pair of HMD and perform the procedure by visualizing the ultrasound images displayed on their HMD screen instead of the ultrasound screen. Each operator will perform an internal jugular vein cannulation via the short-axis approach. Every procedure will be recorded by focusing on the participant's hands and faces.
  Arms: HMD group

SUMMARY:
Head-mounted displays (HMD) in medical practice are current research topics. The goal of this clinical trial is to learn if HMD would improve the safety and efficacy in ultrasound-guided central venous catheterization. The main questions it aims to answer are: Does HMD reduce the procedure time and increase the catheterization success rate in ultrasound-guided central venous catheterization. Does HMD increase the satisfaction score of operators and patients. Researchers will compare HMD with the conventional ultrasound in central venous catheterization. Operators will receive either HMD or conventional ultrasound machine to guide internal jugular vein catheterization. The procedure time, puncture success rate, complication and satisfactory score will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective surgery under general anesthesia
2. Patients indicative of internal jugular vein catheterization.

Exclusion Criteria:

1. A recent history of internal jugular vein puncture, wound, infection, hematomas, nerve injury at the venous cannulation site; 2. Combined with peripheral vascular disease, coagulopathy; 3. History of opiate abuse; 4. Pre-existing chronic pain, mental or neurological disorders; 5. Allergy to local anesthetics or gel; 6. Unstable vital signs, including hypertension, hypotension or arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Total catheterization time | From application of the ultrasound probe to skin to the end of catheterization
  The total catheterization time is defined as the period between the probe positioning on the patient's skin and insertion of the catheter, irrespective of the attempt number of the venous catheterization.

SECONDARY OUTCOMES:
Ultrasound scan time | From application of the ultrasound probe to skin to the end of catheterization
  the time from application of the ultrasound probe to skin to the beginning of puncture
Venous access time | From application of the ultrasound probe to skin to the end of catheterization
  period between skin penetration by the needle and the first flashback of venous blood
Number of needle redirections | From application of the ultrasound probe to skin to the end of catheterization
  the number of times the participant withdraws the needle and re-directs it or advances it at a different angle.
Number of looks at the monitor | From application of the ultrasound probe to skin to the end of catheterization
  The number of times the participant looks at the monitor (ultrasound monitor or head-mounted display) during the procedure based on assessment of the subject's head and eye position noted on video.
Time spent looking at the patient | From application of the ultrasound probe to skin to the end of catheterization
  The total amount of time the patient is the main focal point of the participant's view based on assessment of the subject's head and eye position noted on video.
Time spent looking at the monitor | From application of the ultrasound probe to skin to the end of catheterization
  The total amount of time the participant spends looking at the ultrasound monitor or the head-mounted display based on assessment of the subject's head and eye position noted on video.
First-attempt success rate of internal jugular vein cannulation | From application of the ultrasound probe to skin to the end of catheterization
  The rate of first-attempt success of internal jugular vein cannulation. Successful internal jugular vein cannulation is confirmed by an flashback of venous blood from the catheter.
The second attempt success rate | From application of the ultrasound probe to skin to the end of catheterization
  The rate of second-attempt success of internal jugular vein cannulation. Second-attempt of puncture is defined as the needle withdrawing to the skin and re-puncture.
Number of attempts of needle puncture | From application of the ultrasound probe to skin to the end of catheterization
  number of attempts until successful needle puncture
The incidence and severity of complications | From application of the ultrasound probe to skin to the catheter removal
  The incidence and severity of complications, such as bleeding, hematoma, arrhythmia, nerve injury, arterial puncture, arterial catheterization, failed catheterization, catheter tip malposition, pneumothorax.
pain score of procedure | From application of the ultrasound probe to skin to the end of catheterization
  Patient's pain scale score during the internal jugular vein catheterization
Failure rate of catheterization. | From application of the ultrasound probe to skin to the end of catheterization
  Inability to cannulate the vein in three attempts will be recorded as a failure.
Satisfaction score of patients | From application of the ultrasound probe to skin to the end of catheterization
  Satisfaction score of patients after receiving the total procedure.
Satisfaction score of operators | From application of the ultrasound probe to skin to the end of catheterization
  The operators' satisfaction will be recorded on a 5-point scale, where 1 = worst; 2 = poor; 3 = acceptable; 4 = good; and 5 = best. The questionnaire includes: degree of physical fatigue; degree of visual fatigue; motion sickness or dizziness; willingness to use the device again and to recommend it to colleagues; the contribution to patient management; how easily information was able to be read.
The diameter and depth of the internal jugular vein | From application of the ultrasound probe to skin to the beginning of puncture
  The diameter and depth of the internal jugular vein in the image
Number of attempts of guidewire insertion | From application of the ultrasound probe to skin to the end of catheterization
  number of attempts until successful guidewire insertion
Number of probe repositioning | From application of the ultrasound probe to skin to the end of catheterization
  Number of ultrasound probe repositioning
The distance of tip of the needle from central line of vessel | From application of the ultrasound probe to skin to the end of catheterization
  The distance of tip of the needle from central line of vessel

CONTACTS AND LOCATIONS:
Overall Officials: Ye Zhang, MD, PhD, Study Chair — The Second Hospital of Anhui Medical University
Locations (1):
- Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: 5 years after publication